CLINICAL TRIAL: NCT00949338
Title: A Randomised Trial Comparing The Bladder Volume Consistency Achieved With Two Bladder-Filling Protocols in Prostate Conformal Radiotherapy
Brief Title: Comparing Two Sets of Bladder-Filling Instructions in Treating Patients Undergoing Radiation Therapy For Prostate Cancer. ICORG 05-04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-04 ICORG; ICORG-05-04; EU-20923
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Arm I (Active Comparator): Patients empty their bladders and consume 6 cups of water 30 minutes before undergoing radiotherapy. Patients also undergo bladder volume measurements using a bladder volume instrument (BVI) periodically during treatment.
  Interventions: Procedure: pre-procedural preparation
- Arm II (Experimental): Patients empty their bladders and consume 3 cups of water 30 minutes before undergoing radiotherapy. Patients also undergo bladder volume measurements using a BVI periodically during treatment.
  Interventions: Procedure: pre-procedural preparation

INTERVENTIONS:
Procedure: pre-procedural preparation — Patients empty their bladders and consume 6 cups or 3 cups of water 30 minutes before undergoing radiotherapy.

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Having a full bladder may improve the effectiveness of radiation therapy to the bladder. It is not yet known which set of bladder-filling instructions is more effective in helping patients keep their bladder full during radiation therapy.

PURPOSE: This randomized clinical trial is comparing two sets of bladder-filling instructions in treating patients with prostate cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the consistency in bladder volumes in patients with prostate cancer undergoing conformal radiotherapy, when randomized to one of two sets of bladder-filling instructions.

Secondary

* To compare the incidence of acute and late genitourinary and gastrointestinal toxicity in patients treated with these methods.
* To determine patient satisfaction with the bladder-filling instructions.
* To determine satisfaction of bladder-filling protocols amongst radiation therapists and doctors.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients empty their bladders and consume 6 cups of water 30 minutes before undergoing radiotherapy. Patients also undergo bladder volume measurements using a bladder volume instrument (BVI) periodically during treatment.
* Arm II: Patients empty their bladders and consume 3 cups of water 30 minutes before undergoing radiotherapy. Patients also undergo bladder volume measurements using a BVI periodically during treatment.

In both arms, patients follow their bladder filling instructions and then undergo conformal radiation therapy daily for about 8 weeks.

Patients' perception of symptoms, quality of life, and urinary symptoms are assessed periodically by the International Prostate Symptom Score (I-PSS). Patients' satisfaction with the bladder-filling instructions (i.e., ability to comply with the bladder-filling protocol, the number of incidents of wetting accidents, number of incidents of having to repeat the water drinking on the same day due to machine breakdown or the patient's inability to retain the full bladder for the required amount of time, and the level of frustration) is assessed periodically by the Visual Analogue Scale (VAS).

Staff satisfaction with bladder-filling interventions (i.e., patient compliance with the protocols, acceptance of bladder dose-volume histograms [DVHs], need for re-scan with a fuller bladder, amount of disruption to the therapist's work schedule, number of incidents of wetting accidents, number of incidents of having to repeat the water drinking on the same day due to machine breakdown or the patient's inability to retain the full bladder for the required amount of time, and the level of satisfaction or frustration) is assessed periodically.

After completion of study treatment, patients are followed up periodically for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer
* Undergoing a radical course of radiotherapy

  * Planned treatment in the supine position

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* No history of urinary incontinence or urinary catheterization
* No evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial or if it is felt by the research/medical team that the patient may not be able to comply with the protocol
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No previous surgery for urinary conditions, except transurethral resection of the prostate (TURP)
* Prior transrectal ultrasound (TRUS) allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Consistency of bladder volumes | 2011

SECONDARY OUTCOMES:
Incidence of acute and late genitourinary and gastrointestinal toxicity | 4 years
Patient satisfaction with bladder-filling instructions | 2011
Staff satisfaction of bladder-filling protocols | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, MD, Principal Investigator — Saint Luke's Hospital; John Gerard Armstrong, MD, MB, MRCPI, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Radiation Oncology Network, Dublin, Ireland